CLINICAL TRIAL: NCT00000524
Title: Myocarditis Treatment Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 43; R01HL034744-04 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2013-11

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Myocarditis
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Myocarditis | interventions — Cyclosporine; Prednisone

INTERVENTIONS:
Drug: cyclosporine
Drug: prednisone

SUMMARY:
To determine whether immunosuppressive treatment improved cardiac function in patients with biopsy-proven myocarditis.

DETAILED DESCRIPTION:
BACKGROUND:

Heart failure due to myocarditis can be a devastating illness. At the same time, immunosuppressive therapy is associated with considerable risks of untoward side effects. Clinicians did not know whether, under what circumstances, or in what form, this hazardous treatment should be used in such critically ill patients. In addition, if immunosuppressive therapy was of benefit, then endomyocardial biopsy in patients suspected of having myocarditis was a justified procedure. The trial also provided information concerning the side effects of immuno-suppressive therapy in such patients.

DESIGN NARRATIVE:

Patients were randomized into two treatment arms consisting of conventional therapy alone for congestive heart failure or combined with a twenty-four week regimen of immunosuppressive therapy. Immunosuppressive therapy consisted of prednisone with either cyclosporine or azathioprine. The primary outcome measure was a change in the left ventricular ejection fraction at twenty-eight weeks. Secondary endpoints included survival, failures of therapy, requirements for conventional therapy, assessments of symptoms, myocardial histology, and arrhythmias.

The study completion date listed in this record was obtained from the Query/View/Report (QVR) System.

ELIGIBILITY:
Men and women, 18 years of age or older, with left ventricular failure and biopsy-documented myocarditis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1986-07; Study Completion 1994-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay Mason — University of Utah

REFERENCES:
- [Background] Mason JW, O'Connell JB. Clinical merit of endomyocardial biopsy. Circulation. 1989 May;79(5):971-9. doi: 10.1161/01.cir.79.5.971. PMID 2653662
- [Background] O'Connell JB, Mason JW. Diagnosing and treating active myocarditis. West J Med. 1989 Apr;150(4):431-5. PMID 2660415
- [Background] O'Connell JB, Mason JW. The applicability of results of streamlined trials to clinical practice: the Myocarditis Treatment Trial. Stat Med. 1990 Jan-Feb;9(1-2):193-6; discussion 196-7. doi: 10.1002/sim.4780090126. PMID 2345835
- [Background] Neumann DA, Burek CL, Baughman KL, Rose NR, Herskowitz A. Circulating heart-reactive antibodies in patients with myocarditis or cardiomyopathy. J Am Coll Cardiol. 1990 Nov;16(6):839-46. doi: 10.1016/s0735-1097(10)80331-6. PMID 2229805
- [Background] Mason JW, O'Connell JB, Herskowitz A, Rose NR, McManus BM, Billingham ME, Moon TE. A clinical trial of immunosuppressive therapy for myocarditis. The Myocarditis Treatment Trial Investigators. N Engl J Med. 1995 Aug 3;333(5):269-75. doi: 10.1056/NEJM199508033330501. PMID 7596370
- [Background] Hahn EA, Hartz VL, Moon TE, O'Connell JB, Herskowitz A, McManus BM, Mason JW. The Myocarditis Treatment Trial: design, methods and patients enrollment. Eur Heart J. 1995 Dec;16 Suppl O:162-7. doi: 10.1093/eurheartj/16.suppl_o.162. PMID 8682088